CLINICAL TRIAL: NCT06511622
Title: Impact of Immune Status on Secondary Infections in Patients With Acute Respiratory Failure
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: ARDS-Infectio
Record Dates: First submitted 2024-06-10; First posted 2024-07-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: ARDS
Keywords: ARDS; ECMO; Herpes viridae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective observational study over the period 1/2019 - 02/2024 with the aim of identifying patients with a predisposition to secondary infections.

DETAILED DESCRIPTION:
As a reference center, Charité Universitaetsmedizin Berlin has been treating patients with the most severe form of acute respiratory failure, known as acute respiratory distress syndrome (ARDS), for more than 30 years. Despite lung-protective forms of ventilation and the use of extracorporeal procedures for oxygenation and decarboxylation (ECMO), mortality is around forty percent. In addition to the primary cause of ARDS, further infectious complications often develop during the course of the disease, which delay recovery.

The aim of this study is to investigate infectious complications (ventilator-associated pneumonia, reactivation of Herpes viridae, pathogen resistance despite formally correct therapy, fungal infections) depending on the immune status.

ELIGIBILITY:
Inclusion Criteria:

* Male and female acute respiratory distress syndrome patients who had an immune status within 48 h of admission
* Patients who received intensive care treatment for acute respiratory distress syndrome ward 8i at Charité in the period from 01/2019 to 02/2024 with a maximum follow-up period of 90 days

Exclusion Criteria:

* None

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients who received intensive care treatment for acute respiratory distress syndrome on ward 8i at Charité in the period from 01/2019 to 02/2024 with a maximum follow-up period of 90 days.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Herpes simplex reactivation | 01/2019- 12/2025
  semi-quantitatively with Herpes simplex (negative / slightly positive / positive and strongly positive) in blood or bronchial lavage
Cytomegalovirus reactivation | 01/2019- 12/2025
  as absolute copy number per milliliter of blood or bronchioalveolar lavage
Epstein Barr virus reactivation | 01/2019- 12/2025
  absolute copy number per milliliter of blood or bronchioalveolar lavage
B cells (CD19 positive) | 01/2019- 12/2025
  Absolute number per nanoliter and percentage of lymphocytes
Natural killer cells Cells (CD16 pos) | 01/2019- 12/2025
  Absolute number per nanoliter and percentage of lymphocytes.
T helper cells (CD4) | 01/2019- 12/2025
  Aabsolute number per nanoliter and percentage of lymphocytes
Cytotoxic T cells (CD8) | 01/2019- 12/2025
  Absolute number per nanoliter and percentage of lymphocytes
HLA-DR expression on monocytes | 01/2019- 12/2025
  in molecules per cell

SECONDARY OUTCOMES:
Beginn weaning | 01/2019- 12/2025
  Days until the first successful spontaneous breathing trial.
Extracorporeal membrane oxygenation duration | 01/2019- 12/2025
  Extracorporeal membrane oxygenation is measured in days
Costs of treatment | 01/2019- 12/2025
  Costs of treatment are measured by costs of particular microbiological diagnostics and therapy.
Pathogen persistence after guideline-compliant therapy (yes/no) | 01/2019- 12/2025
Ventilator-associated pneumonia (yes/no) | 01/2019- 12/2025
Occurrence of fungal pneumonia (yes/no) | 01/2019- 12/2025
Mortality | 01/2019- 12/2025
  ITS mortality and hospital mortality are measured.
Sequential Organ Failure Assessment (SOFA score) | 01/2019- 12/2025
  Routine patient treatment data - score is measured numerically (0 - 24) Routine patient treatment data.
Simplified Acute Physiology Score (SAPS II) | 01/2019- 12/2025
  Routine patient treatment data - score is measured numerically (0 - 163)
Pre-existing conditions | 01/2019- 12/2025
  Classified recording of previous illnesses (e.g. haematological diseases, tumour diseases, chronic heart failure, etc.) from the medical file.
Concomitant infections with therapy | 01/2019- 12/2025
  Results of microbiological diagnostics (growth- and molecular-based diagnostics) by specifying the name of the pathogen.
Volumes | 01/2019- 12/2025
  Volumes administered, incl. transfusions and coagulation factors
Ventilation parameters | 01/2019- 12/2025
  Recording of ventilation parameters such as airway, ventilation mode and start of ventilation weaning.
Catecholamine doses | 01/2019- 12/2025
  Name of catecholamines, inotropes and vasopressors
Number of catecholamine days | 01/2019- 12/2025
  Number of days with dose of norepinephrine > 0.1 µg/kg/min for more than 30 min or equivalent dose of other catecholamines.
Recording of end organ damage such as liver and kidney failure | 01/2019- 12/2025
  Organ damage measured by routine laboratory
Diagnoses during the intensive care stay | 01/2019- 12/2025
  Diagnoses as the cause of ARDS, but also newly acquired diagnoses such as critical illness myopathy / polyneuropathy, renal failure.
Administration of immunosuppressants | 01/2019- 12/2025
  Administration of immunosuppressants like corticosteroid, chemotherapy, monoclonal antibodies within the last 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No